CLINICAL TRIAL: NCT04410237
Title: Triamcinolone Acetonide Injections in Mild-to-moderate Chronic Plaque Psoriasis With a Novel Needle-free Drug-delivery System: an Observational Pilot Study
Brief Title: Triamcinolone Acetonide Injections in Mild-to-moderate Chronic Plaque Psoriasis With a Novel Needle-free Drug-delivery System
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Neil Korman, Principle Investigator, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY20200508
Record Dates: First submitted 2020-05-20; First posted 2020-06-01 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Psoriasis
Keywords: Triamcinolone Acetonide; Med-Jet
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Med-Jet (Experimental): The Med-Jet injector is a novel needle-free drug-delivery system, which we believe may be a solution to the impracticalities of ILTA for mild-to-moderate psoriasis. It uses regulated compressed air as a power source to accelerate an injectable fluid through a 0.005" orifice (6x smaller than a 30G needle) to penetrate the skin and deliver medication to a specific anatomical region.12 The drug-delivery device is highly configurable allowing adjustable depth and volume parameters.12 In addition, the high-performance design allows for triggering multiple injection sites rapidly which is practical when needing to treat large surface areas
  Interventions: Device: Med-Jet
- Traditional Syringe (Active Comparator): TAC will be injected on a half-plaque while the control half of the plaque will be untreated. A standard sterile disposable 1 ml syringe and 30-gauge needle will be used to inject TAC.
  Interventions: Other: Traditional Syringe

INTERVENTIONS:
Device: Med-Jet — One half of each psoriasis plaque will be treated with a Med-Jet device and Triamcinolone acetonide (TAC) while the control half will be untreated.
  One side of the body will be treated using a conventional syringe and the opposite side of the body will be treated using the Med-Jet needle-free injection device to verify efficacy, safety, and pain score
  Arms: Med-Jet
Other: Traditional Syringe — One half of each psoriasis plaque will be treated with a traditional syringe and Triamcinolone acetonide (TAC) while the control half will be untreated.
  One side of the body will be treated using conventional syringe and the opposite side of the body will be treated using the Med-Jet needle-free injection device to verify efficacy, safety, and pain score
  Arms: Traditional Syringe

SUMMARY:
This is an observational pilot study comparing triamcinolone acetonide injections with the investigational Med-jet needle-free drug-delivery system as an alternative to using a conventional syringe and needle in patients with mild-to-moderate psoriasis. There will be five (5) visits necessary for study participation. The hypothesis is that the efficacy, safety, pain tolerance, and quality of life (QoL) metrics of the Med-jet needle-free drug-delivery system will be equal to or superior to that of a conventional syringe and needle.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with plaque-type psoriasis defined by either:

  * A board-certified dermatologist, OR
  * Dermatology Nurse Practitioner, OR
  * Skin punch biopsy
* Involvement of body surface area (BSA) < 10% at screening and baseline visit.
* The presence of plaque-type psoriasis at least two (2) plaques that are at least two (2) cm² in areas of the trunk, buttock, or extremities that are either:

  * Symmetrically located on contralateral body site OR
  * Within the same body site but separated by ≥ 1 cm
* Able to give informed consent under IRB approval procedures

Exclusion Criteria:

* Known allergy or hypersensitivity to triamcinolone acetonide
* Pregnant, breastfeeding, or planning to get pregnant 4 weeks before, during, and 4 weeks after the study.
* Inability to provide informed consent
* Active untreated diseases or medication usage which may interfere with wound healing and immune function (anti-neoplastic, systemic immunosuppressants, anticoagulants, daily NSAIDS)
* Use of tanning booths for at least 4 weeks prior to baseline visit
* Current or recent use of topical steroid, tar, phototherapy, Vitamin D, or retinoid therapy to target lesions for at least 2 weeks prior to baseline visit
* Current or recent use of systemic or biologic therapy for at least 4 weeks or 5 half-lives of the drug (whichever is longer) prior to baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCASE v5.0 | 26 Weeks
  Validate the safety of the Med-jet needle-free drug-delivery system in combination with triamcinolone acetonide in patients with mild-to-moderate psoriasis.

SECONDARY OUTCOMES:
Efficacy as measured by the target physician global assessment | 26 Weeks
  Validate efficacy as alternatives to using triamcinolone acetonide with a conventional needle and syringe in patients with mild-to-moderate psoriasis as measured by the target physician global assessment (tPGA). tPGA is a 5 point scale (0-4) 0 meaning clear skin and 4 meaning severe skin.
Tolerability as measured by the visual analog pain scores | 26 Weeks
  Validate tolerability as alternatives to using triamcinolone acetonide with a conventional needle and syringe in patients with mild-to-moderate psoriasis as measured by the visual analog pain scores. Measured on a scale of 0 to 10, where 0 is no distress and 10 is unbearable distress.
Quality of Life metric as assessed by the dermatology life quality assessment | 26 Weeks
  Validate quality of life metrics as alternatives to using triamcinolone acetonide with a conventional needle and syringe in patients with mild-to-moderate psoriasis as measured by the dermatology life quality assessment (DLQI). DLQI is 0 to 30 scale, where 0 is no effect on patient life and 30 is an extremely large effect on patient life.
Pruritus as measured by visual analog pruritus scale | 26 weeks
  Validate pruritus as alternatives to using triamcinolone acetonide with a conventional needle and syringe in patients with mild-to-moderate psoriasis as measured by the visual analog pruritus scale, measured on a scale of 0 to 10 where 0 is no itch and 10 is the worst itch imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Korman, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gelfand JM, Stern RS, Nijsten T, Feldman SR, Thomas J, Kist J, Rolstad T, Margolis DJ. The prevalence of psoriasis in African Americans: results from a population-based study. J Am Acad Dermatol. 2005 Jan;52(1):23-6. doi: 10.1016/j.jaad.2004.07.045. PMID 15627076
- [Background] Parisi R, Symmons DP, Griffiths CE, Ashcroft DM; Identification and Management of Psoriasis and Associated ComorbidiTy (IMPACT) project team. Global epidemiology of psoriasis: a systematic review of incidence and prevalence. J Invest Dermatol. 2013 Feb;133(2):377-85. doi: 10.1038/jid.2012.339. Epub 2012 Sep 27. PMID 23014338
- [Background] Yeung H, Takeshita J, Mehta NN, Kimmel SE, Ogdie A, Margolis DJ, Shin DB, Attor R, Troxel AB, Gelfand JM. Psoriasis severity and the prevalence of major medical comorbidity: a population-based study. JAMA Dermatol. 2013 Oct;149(10):1173-9. doi: 10.1001/jamadermatol.2013.5015. PMID 23925466
- [Background] Stern RS, Nijsten T, Feldman SR, Margolis DJ, Rolstad T. Psoriasis is common, carries a substantial burden even when not extensive, and is associated with widespread treatment dissatisfaction. J Investig Dermatol Symp Proc. 2004 Mar;9(2):136-9. doi: 10.1046/j.1087-0024.2003.09102.x. PMID 15083780
- [Background] Fouere S, Adjadj L, Pawin H. How patients experience psoriasis: results from a European survey. J Eur Acad Dermatol Venereol. 2005 Nov;19 Suppl 3:2-6. doi: 10.1111/j.1468-3083.2005.01329.x. PMID 16274404
- [Background] Alinia H, Moradi Tuchayi S, Smith JA, Richardson IM, Bahrami N, Jaros SC, Sandoval LF, Farhangian ME, Anderson KL, Huang KE, Feldman SR. Long-term adherence to topical psoriasis treatment can be abysmal: a 1-year randomized intervention study using objective electronic adherence monitoring. Br J Dermatol. 2017 Mar;176(3):759-764. doi: 10.1111/bjd.15085. Epub 2016 Nov 29. PMID 27664969
- [Background] Kamel JG, Yamauchi PS. Managing Mild-to-Moderate Psoriasis in Elderly Patients: Role of Topical Treatments. Drugs Aging. 2017 Aug;34(8):583-588. doi: 10.1007/s40266-017-0480-8. PMID 28755089
- [Background] READETT MD. Intralesional triamcinolone acetonide in the treatment of psoriasis. Br J Dermatol. 1961 Mar;73:107-9. doi: 10.1111/j.1365-2133.1961.tb14416.x. No abstract available. PMID 13740078
- [Background] HASEGAWA J, LIVINGSTON W. The intralesional use of triamcinolone acetonide in psoriasis. A double blind study. Arch Dermatol. 1962 Feb;85:258-60. doi: 10.1001/archderm.1962.01590020098010. No abstract available. PMID 13905149
- [Background] WEIDMAN AI. Treatment of psoriasis and other dermatoses with intralesional injections of triamcinolone acetonide. Curr Ther Res Clin Exp. 1963 Jan;5:7-11. No abstract available. PMID 13999537
- [Background] McLenon J, Rogers MAM. The fear of needles: A systematic review and meta-analysis. J Adv Nurs. 2019 Jan;75(1):30-42. doi: 10.1111/jan.13818. Epub 2018 Sep 11. PMID 30109720
- [Background] PARISER H, MURRAY PF. Intralesional injections of triamcinolone. Effects of different concentrations on psoriatic lesions. Arch Dermatol. 1963 Feb;87:183-7. doi: 10.1001/archderm.1963.01590140045008. No abstract available. PMID 13941443
- [Background] Schramm-Baxter JR, Mitragotri S. Investigations of needle-free jet injections. Conf Proc IEEE Eng Med Biol Soc. 2004;2004:3543-6. doi: 10.1109/IEMBS.2004.1403996. PMID 17271055
- [Background] Park G, Modak A, Hogan NC, Hunter IW. The effect of jet shape on jet injection. Annu Int Conf IEEE Eng Med Biol Soc. 2015;2015:7350-3. doi: 10.1109/EMBC.2015.7320089. PMID 26737989
- [Background] Vadeboncoeur S, Richer V, Nantel-Battista M, Benohanian A. Treatment of Palmar Hyperhidrosis With Needle Injection Versus Low-Pressure Needle-Free Jet Injection of OnabotulinumtoxinA: An Open-Label Prospective Study. Dermatol Surg. 2017 Feb;43(2):264-269. doi: 10.1097/DSS.0000000000000970. PMID 27893541
- [Background] Nantel-Battista M, Richer V, Marcil I, Benohanian A. Treatment of nail psoriasis with intralesional triamcinolone acetonide using a needle-free jet injector: a prospective trial. J Cutan Med Surg. 2014 Jan-Feb;18(1):38-42. doi: 10.2310/7750.2013.13078. PMID 24377472